CLINICAL TRIAL: NCT00002976
Title: A Randomized Double-Blinded Trial of Estrogen Replacement Therapy Versus Placebo in Women With Stage I or II Endometrial Adenocarcinoma
Brief Title: Estrogen Replacement Therapy in Treating Women With Early-Stage Endometrial Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Eastern Cooperative Oncology Group (Network); SWOG Cancer Research Network (Network)
Organization: GOG Foundation (Network)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000065498; GOG-137A; E-G0137; SWOG-G0137
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2003-04

CONDITIONS: Endometrial Cancer
Keywords: stage I endometrial carcinoma; stage II endometrial carcinoma; endometrial adenocarcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Estrogens, Conjugated (USP)

INTERVENTIONS:
Drug: conjugated estrogens

SUMMARY:
RATIONALE: Estrogen replacement therapy may improve quality-of-life in postmenopausal women with endometrial cancer. It is not yet known whether estrogen replacement therapy will affect cancer recurrence.

PURPOSE: Randomized double-blinded phase III trial to determine the effectiveness of estrogen replacement therapy in treating women who have stage I or stage II endometrial cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the effect of estrogen replacement therapy on recurrence free and overall survival in women with a history of stage I or II endometrial adenocarcinoma.

OUTLINE: This is a randomized, double blind study. Patients are stratified according to stage of endometrial cancer (IA vs IB/IC vs II). Patients are randomized to one of two treatment arms:

* Arm I: Patients receive oral conjugated estrogens (Premarin) daily for 3 years.
* Arm II: Patients receive oral placebo daily for 3 years. Patients are followed every 6 months for 3 years and then annually for 2 years.

PROJECTED ACCRUAL: Approximately 2,108 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed grade I, II or III endometrial adenocarcinoma (endometrioid, villoglandular, mucinous, adenosquamous, papillary serous, clear cell, or not otherwise specified)
* Must have had total hysterectomy and bilateral salpingo-oophorectomy within past 20 weeks

  * Surgical stage IA, IB, IC, IIA (occult), or IIB (occult) disease
* Must have had normal mammogram, or a negative breast biopsy after an abnormal mammogram, within past year

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin no greater than 1.5 times normal
* SGOT no greater than 3 times normal
* No acute liver disease

Renal:

* Not specified

Cardiovascular:

* No prior thromboembolic disease

Other:

* No prior or current carcinoma of the breast
* No other prior invasive malignancy within the past 5 years except nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* No concurrent hormonal therapy

Radiotherapy:

* Not specified

Surgery:

* See Disease Characteristics
* Recovered from prior surgery

Other:

* No prior cancer treatment that would preclude study therapy
* Concurrent participation on GOG Lap-1 or GOG Lap-2 allowed

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2108 (Estimated)
Dates: Start 1997-06; Primary Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard R. Barakat, MD, Study Chair — Memorial Sloan Kettering Cancer Center; Scott Wadler, MD, Study Chair — Albert Einstein College of Medicine; David S. Alberts, MD, Study Chair — University of Arizona
Locations (149):
- United States (149):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Carl T. Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock (McClellan), Little Rock, Arkansas
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Veterans Affairs Medical Center - West Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Community Hospital of Los Gatos, Los Gatos, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Medical Center, Sacramento, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - New Britain, Connecticut
  - MBCCOP-Howard University Cancer Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Mayo Clinic, Jacksonville, Florida
  - Sacred Heart Hospital of Pensacola, Pensacola, Florida
  - Tampa Bay Cancer Consortium, St. Petersburg, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Medical College of Georgia Comprehensive Cancer Center, Savannah, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - Earl K. Long Medical Center, Baton Rouge, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Ochsner Clinic, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Butterworth Hospital, Grand Rapids, Michigan
  - CCOP - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Beaumont, Royal Oak, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Biloxi, Biloxi, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Department of OB-GYN, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Methodist Cancer Center - Omaha, Omaha, Nebraska
  - Cooper Hospital/University Medical Center, Camden, New Jersey
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Cancer Center of Albany Medical Center, Albany, New York
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - Crouse Hospital, Syracuse, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Southern Pines Women's Health Center, Southern Pines, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - University of Tennessee Cancer Institute, Winston-Salem, North Carolina
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Barrett Cancer Center, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Oklahoma City, Oklahoma City, Oklahoma
  - University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - Good Samaritan Hospital Comprehensive Cancer Center, Portland, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - OHSU Cancer Institute, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - Veterans Affairs Medical Center - Charleston, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - Baptist Regional Cancer Center - Knoxville, Knoxville, Tennessee
  - University of Tennessee Medical Center at Knoxville, Knoxville, Tennessee
  - Brookview Research, Inc., Nashville, Tennessee
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - CCOP - M.D. Anderson Research Base, Houston, Texas
  - Covenant Health System, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - Fletcher Allen Health Care - Medical Center Campus, Burlington, Vermont
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - Eastern Virginia Medical School, Norfolk, Virginia
  - Massey Cancer Center, Richmond, Virginia
  - University of Virginia at Roanoke, Roanoke, Virginia
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin

REFERENCES:
- [Result] Barakat RR, Bundy BN, Spirtos NM, Bell J, Mannel RS; Gynecologic Oncology Group Study. Randomized double-blind trial of estrogen replacement therapy versus placebo in stage I or II endometrial cancer: a Gynecologic Oncology Group Study. J Clin Oncol. 2006 Feb 1;24(4):587-92. doi: 10.1200/JCO.2005.02.8464. PMID 16446331